CLINICAL TRIAL: NCT00757640
Title: The CHOLEGAS Study: Multicentric Randomized, Double-blinded, Controlled Trial of Gastrectomy Plus Prophylactic Cholecystectomy Versus Gastrectomy Only, in Adults Submitted to Gastric Cancer Surgery With Curative Intent.
Brief Title: Gastrectomy Plus Prophylactic Cholecystectomy in Gastric Cancer Surgery
Acronym: CHOLEGAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Italian Research Group for Gastric Cancer (Network)
Collaborators: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Bencini Lapo, Dr, PhD, Italian Research Group for Gastric Cancer
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Firenze 1
Record Dates: First submitted 2008-09-20; First posted 2008-09-23 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, surgery, prophylactic cholecystectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Cholecystectomy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (No Intervention): no cholecystectomy
- A (Experimental): cholecystectomy
  Interventions: Procedure: cholecystectomy

INTERVENTIONS:
Procedure: cholecystectomy — prophylactic cholecystectomy during standard gastric surgery for cancer
  Arms: A

SUMMARY:
The patients will be divided into two groups: in the first group the patient will be submitted to prophylactic cholecystectomy during standard surgery for curable gastric cancer (subtotal or total gastrectomy), while in the second group will be submitted to standard gastric surgery only.

DETAILED DESCRIPTION:
The incidence of gallstones and gallbladder sludge is known to be higher in patients after gastrectomy than in general population. This higher incidence is probably related to surgical dissection of the vagus nerve branches and the anatomical gastrointestinal reconstruction. Therefore, some surgeons perform routine concomitant cholecystectomy during standard surgery for gastric malignancies. However, not all the patients who are diagnosed to have cholelithiasis after gastric cancer surgery will develop symptoms or require additional surgical treatments and a standard laparoscopic cholecystectomy is feasible even in those patients who underwent previous gastric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing standard gastric surgery for cancer

Exclusion Criteria:

* gallbladder disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Reduced biliary complications | 5 years

SECONDARY OUTCOMES:
Improved quality of life | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Marco Farsi, MD, Principal Investigator — Chirurgia Generale e Oncologica Azienda Ospedaliero-Universitaria Careggi
Locations (1):
- Azienda Ospedaliero-Universitaria Careggi - Chirurgia Generale ed Oncologica, Florence, Italy

REFERENCES:
- [Derived] Bernini M, Bencini L, Sacchetti R, Marchet A, Cristadoro L, Pacelli F, Berardi S, Doglietto GB, Rosa F, Verlato G, Cozzaglio L, Bechi P, Marrelli D, Roviello F, Farsi M; Italian Research Group for Gastric Cancer (IRGGC). The Cholegas Study: safety of prophylactic cholecystectomy during gastrectomy for cancer: preliminary results of a multicentric randomized clinical trial. Gastric Cancer. 2013 Jul;16(3):370-6. doi: 10.1007/s10120-012-0195-9. Epub 2012 Sep 5. PMID 22948317
- [Derived] Farsi M, Bernini M, Bencini L, Miranda E, Manetti R, de Manzoni G, Verlato G, Marrelli D, Pedrazzani C, Roviello F, Marchet A, Cristadoro L, Gerard L, Moretti R; GIRCG (Gruppo Italiano di Ricerca sul Cancro Gastrico). The CHOLEGAS study: multicentric randomized, blinded, controlled trial of gastrectomy plus prophylactic cholecystectomy versus gastrectomy only, in adults submitted to gastric cancer surgery with curative intent. Trials. 2009 May 15;10:32. doi: 10.1186/1745-6215-10-32. PMID 19445661
- See also: official site of group study — http://www.gircg.it/